CLINICAL TRIAL: NCT06922721
Title: ATICC: A Mixed-Methods Study on Addiction, Trauma, and Immigration Among Vulnerable Young Adults in the Grand Est Youth Network
Brief Title: Protocol Study on Addiction, Trauma and Immigration Among Vulnerable Young Adults in Grand Est
Acronym: ATICC
Status: Recruiting | Type: Observational
Sponsor: University of Lorraine (Other)
Collaborators: French Institute for Public Health Research (IReSP) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024-A01534-43
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Trauma and Stress-related Disorders; Substance Use Disorder (SUD); Substance Use Risk
Keywords: addiction; trauma; Immigration; Mental health; young adults; Substance use
MeSH Terms: conditions — Trauma and Stressor Related Disorders; Substance-Related Disorders; Behavior, Addictive; Wounds and Injuries; Psychological Well-Being | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- group participants: Participant aged >18, Resident in a Housing center , Fluent in French, adult participants who are not under guardianship (tutelle) or curatorship (curatelle).
  Interventions: Other: Focus group

INTERVENTIONS:
Other: Focus group — The "Well-Being Coffee Group" intervention is implemented in two formats: in person and others via videoconference, all facilitated by the same psychologist throughout the study. Across all formats, participation is voluntary and follows an information phase and the signing of an informed consent form. Participants will complete standardized evaluation questionnaires at multiple time points. The discussion groups are designed to create a supportive and open environment that encourages free expression. Their goal is to provide participants with a space to share their thoughts, emotions, and personal experiences, as well as to reflect on those emerging from group discussions. Topics explored include identity, substance use, migratory experiences, and mental health, fostering meaningful dialogue and mutual support.

SUMMARY:
The ATICC study (Addiction, Trauma, and Immigration, Prevention and Cross-Cultural Support for Care) investigates the complex relationships between trauma, substance use, migration experiences, and mental health perceptions among vulnerable young adults in Transitional Housing (Foyers de Jeunes Travailleurs) in France. Using a tripartite methodology, the study includes: (1) a cross-sectional survey to identify risk factors, (2) qualitative interviews to explore individual experiences, and (3) a longitudinal intervention using focus groups to assess psychological well-being and attitudes toward care. The findings will contribute to developing culturally adapted prevention and support programs.

DETAILED DESCRIPTION:
The ATICC study (Addiction, Trauma, and Immigration, Prevention and Cross-Cultural Support for Care) is a mixed-methods research project aimed at understanding the interplay between trauma, substance use, migration experiences, and mental health perceptions among vulnerable young adults residing in Transitional Housing for Young Adults (Foyers de Jeunes Travailleurs, FJT) in France. The study will identify key risk factors, assess barriers to healthcare access, and evaluate the effectiveness of group interventions in improving psychological well-being and attitudes toward mental health services.

The study is structured into three complementary research components:

Cross-sectional study: Utilizes standardized questionnaires to assess substance use behaviors, trauma history, mental health status, and barriers to healthcare. The data will be collected at baseline and analyzed using descriptive and multivariate statistical techniques (R software).

Qualitative study: Conducts semi-structured interviews with a subset of participants who engage in substance use. Thematic analysis using NVivo software will be applied to explore individual narratives and subjective experiences related to substance use and mental health perceptions.

Longitudinal interventional study: Implements focus group interventions within transitional housing settings to evaluate their impact on psychological well-being and attitudes toward healthcare. Pre- and post-intervention assessments will be conducted using validated psychological measures.

Data will be analyzed using mixed models and appropriate statistical corrections to assess intervention effectiveness.

Registry procedures and quality factors include a Quality Assurance Plan ensuring data validation, site monitoring, and ethical compliance through adherence to the Committee for the Protection of Persons (CPP) Ile-de-France; Data Checks & Source Data Verification through automated validation rules and cross-checking against medical records; a Data Dictionary defining all variables, including sources, coding systems (e.g., ICD-10, WHO Drug Dictionary, MedDRA), and reference ranges; and Standard Operating Procedures (SOPs) for participant recruitment, data collection, data management, adverse event reporting, and change management to ensure consistency and compliance. The Sample Size Assessment includes at least 300 participants for the cross-sectional study to ensure statistical power, 40 participants for qualitative interviews to achieve data saturation, and 6-8 participants per focus group session, with repeated measures over six months to track changes. The plan for Missing Data incorporates multiple imputation techniques, sensitivity analyses, and data inconsistency reviews. The statistical analysis plan includes descriptive analyses for mean, median, and standard deviations, and inferential analyses using logistic regression for risk factor identification, mixed-effects models for intervention outcomes, and thematic coding for qualitative data analyzed with NVivo software. Ethical considerations and registration details confirm that the study has received ethical approval from the CPP Ile-de-France (November 18, 2024) and is registered with the French National Agency for the Safety of Medicines and Health Products (ANSM) under ID-RCB: 2024-A01534-43, with participant confidentiality maintained through anonymized data storage and GDPR-compliant procedures. This detailed description provides the necessary technical information on the ATICC study, ensuring compliance with clinical trial registration requirements.

ELIGIBILITY:
Inclusion Criteria:

* Resident in a Housing center, speak and read french, adult participants who are not under guardianship or curatorship, any cultural background.

Exclusion Criteria:

* minors, don't speak and read french, adults under guardianship and curatorship.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of young adults aged 16 to 25 years residing in Transitional Housing for Young Adults (Foyers de Jeunes Travailleurs, FJT) affiliated with the Union Régionale pour l'Habitat des Jeunes (URHAJ). These individuals meet specific vulnerability criteria and come from diverse life trajectories, including those aging out of child welfare services (ASE), individuals under judicial protection (PJJ), persons with disabilities, refugees, and single-parent families. Due to their backgrounds, these young adults face significant adversity, which may have profound effects on their mental health and well-being. This population is particularly exposed to psychosocial stressors, making them a relevant demographic for studying the interplay between trauma, substance use, and mental health care access.
Sampling Method: Non-Probability Sample
Enrollment: 182 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Attitudes toward mental health care | 6 months
  Attitudes toward mental health care is measured through changes in perceptions of mental health services, stigma, and willingness to seek care before and after the intervention through a validated scale.

SECONDARY OUTCOMES:
Anxiety | 6 months
  Anxiety is a mental health condition characterized by excessive worry, fear, or nervousness that can interfere with daily functioning. Generalized Anxiety Disorder (GAD) is one of the most common forms assessed using the GAD-7, a self-report screening measure developed to address limitations in existing anxiety assessments. The GAD-7, consisting of seven questions, is widely used in adult primary care and psychiatric settings due to its efficiency, reliability, and sensitivity to treatment-related changes.
Depression | 6 months
  Depression is a mood disorder characterized by persistent sadness, loss of interest or pleasure in activities, and other symptoms that interfere with daily life. It can vary in severity and last for weeks, months, or even years. Depression in this study will be assessed using the PHQ-9, a screening tool used to assess the presence and severity of depression. It is based on the nine diagnostic criteria for major depressive disorder from the DSM-IV. Each question in the PHQ-9 assesses a specific symptom of depression and is rated on a scale from 0 to 3, depending on how often the symptom has been experienced in the last two weeks.
Alcohol use | 6 months
  Alcohol use will be assessed using the Alcohol Use Disorders Identification Test (AUDIT) to identify individuals with risky or harmful alcohol consumption and detect alcohol dependence.
  The AUDIT questionnaire consists of 10 questions, divided into three categories, alcohol consumption, alcohol-Related problems and signs of alcohol dependence.
Tobacco use | 6 months
  Nicotine dependence is going to be assessed the Fagerström test for nicotine dependence that measures the level of nicotine addiction in individuals who smoke cigarettes. Each question is designed to evaluate the degree of nicotine dependence based on smoking behaviors.
Cannabis use | 6 months
  Cannabis Abuse Screening Test (CAST) will be used to assess cannabis consumption. It is a six-question tool used to assess problematic cannabis use, and evaluates behaviors linked to cannabis use disorder (CUD), such as frequent consumption, inability to control use, neglect of responsibilities, tolerance, withdrawal symptoms, and continued use despite negative consequences.

CONTACTS AND LOCATIONS:
Overall Officials: Aziz Essadek, Phd in psychology, Study Director — University of Lorraine
Locations (7):
- France (7):
  - Les Compagnons du Devoir et du Tour de France, Jarville-la-Malgrange
  - Résidence Habitat Jeunes Campus, Maxéville
  - Association Carrefour, Metz
  - Foyer des jeunes ouvriers, Metz
  - Résidence des Abeilles ADALI-HABITAT, Nancy
  - Résidence MARAE, Nancy
  - Habitat Jeunes 3 frontières, Thionville

IPD SHARING:
Plan to Share IPD: No
We will not share individual participant data (IPD) in order to protect the privacy and confidentiality of our study participants. Our publications will present aggregate findings and summary statistics without revealing any identifiable details.

REFERENCES:
- [Derived] Najdini M, Frigaux A, Mathieu J, Shadili G, Guenoun T, Vlachopoulou X, Belot RA, Bazan A, Gressier F, Robin M, Essadek A. ATICC: a mixed-methods study on addiction, trauma, and immigration among vulnerable young adults in the grand est youth network. BMC Psychol. 2025 May 30;13(1):582. doi: 10.1186/s40359-025-02738-5. PMID 40448223
- See also: Related Info — https://interpsy.univ-lorraine.fr/aticc/